CLINICAL TRIAL: NCT05607927
Title: Laparoscopic Proximally Extended Colorectal Resection With Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Late Complications of Chronic Radiation-induced Rectal Injury: A Prospective, Multicenter, Randomized Controlled Clinical Trail
Brief Title: PE-Bacon for Late Complications of Chronic Radiation-induced Rectal Injury
Acronym: PE-Bacon
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE-Bacon2022
Record Dates: First submitted 2022-09-26; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Chronic Radiation Injury
Keywords: PE-Bacon; Parks; complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parks surgery group (Other): The CRII patients received Parks surgery
  Interventions: Procedure: Parks surgery
- PE-Bacon surgery group (Experimental): The CRII patients received PE-Bacon surgery
  Interventions: Procedure: PE-Bacon surgery

INTERVENTIONS:
Procedure: Parks surgery — Parks surgery
  Arms: Parks surgery group
Procedure: PE-Bacon surgery — PE-Bacon surgery
  Arms: PE-Bacon surgery group

SUMMARY:
Chronic radiation-induced injury (CRII) is a common complication after radiation therapy for pelvic malignancies. Resection surgery could be an optimal surgical approach when CRII is complicated by late complications. However, because of high incidence of postoperative complications like anastomotic leakage rate and mortality, doctors try to avoid performing surgical resection. In addition, there is sparse agreement on the types of surgery.

Previous study proved that anastomosis with at least one end of bowel without radiation damage can greatly reduce postoperative anastomotic leakage rate and mortality. And in Bacon surgery, primary anastomosis is not performed, and the anastomotic tension markedly reduced and the blood supply of anastomosis can be judged intuitively to improve the quality of anastomosis in the second stage of intestinal anastomosis to decrease the anastomotic leakage rate. Combining the advantages of proximally extended resection and two-stage anastomosis could minimize potential complications and maximize the therapeutic efficacy in theory, and a small sample prospective clinical study by the investigator have already preliminarily confirmed it. The investigator has also preliminarily proved that Parks surgery is safe and feasible for the treatment of late complications of CRII.

Therefore, this study aims to observe the safety and effectiveness of PE-Bacon surgery with Parks surgery as a control, in order to select more optimal surgical methods and provide a high-level evidence-based medical basis for patients with late complications of CRII.

DETAILED DESCRIPTION:
Chronic radiation-induced injury (CRII) is a common complication after radiation therapy for pelvic malignancies. Compared with diversion surgery, resection surgery removes the damaged tissue completely to avoid the risks of recurrence and improve patients' outcome. Hence, resection surgery could be an optimal surgical approach when CRII is complicated by late complications. However, because of high incidence of postoperative complications like anastomotic leakage rate and mortality, doctors try to avoid performing surgical resection. In addition, there is sparse agreement on the types of surgery.

With the advances of surgical techniques and perioperative care, the morbidity and mortality of resection surgery has been decreased significantly. In addition, previous study proved that anastomosis with at least one end of bowel without radiation damage can greatly reduce postoperative anastomotic leakage rate and mortality. And in Bacon surgery, primary anastomosis is not performed, and the anastomotic tension markedly reduced and the blood supply of anastomosis can be judged intuitively to improve the quality of anastomosis in the second stage of intestinal anastomosis to decrease the anastomotic leakage rate. Combining the advantages of proximally extended resection and two-stage anastomosis could minimize potential complications and maximize the therapeutic efficacy in theory, and a small sample prospective clinical study by the investigator have already preliminarily confirmed it. And the investigator has also preliminarily proved that Parks surgery is safe and feasible for the treatment of late complications of CRII.

Therefore, this study aims to observe the safety and effectiveness of PE-Bacon surgery with Parks surgery as a control, in order to select more optimal surgical methods and provide a high-level evidence-based medical basis for patients with late complications of CRII.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-70 years;
* 2. Patients with Eastern Cooperative Oncology Group (ECOG) physical condition score of 0-2;
* 3. Patients with previous pathological diagnosis of pelvic tumors (Gynecology, prostate, urinary system);
* 4. Patients with a history of pelvic radiotherapy, at least 6 months from the end of the last radiotherapy;
* 5. Patients without recurrence or metastasis of primary tumor;
* 6. The late complications of CRII patients, such as deep rectal ulcer (VRS score >=3), rectal sigmoid colon stenosis, obstruction, chronic perforation, rectal necrosis, rectovaginal fistula, intractable anal pain caused by rectal lesions, intractable rectal bleeding which is still difficult to be relieved by stoma operation, and patients who need sigmoid colorectal resection;
* 7. Patients who can tolerate general anesthesia;
* 8. The subjects and their families are able to understand the study plan, willing to participate and sign the informed consent.

Exclusion Criteria:

* 1. Patients with acute intestinal obstruction, acute intestinal perforation and intestinal hemorrhage who need emergency operation;
* 2. Patients with severe pelvic adhesion and frozen pelvis;
* 3. Patients with unstable primary tumor or tumor in other parts;
* 4. Patients who need to undergo combined organ resection;
* 5. Patients with a history of sigmoidostomy;
* 6. American society of anesthesiologists (ASA) level IV to V;
* 7. Patients with serious mental illness;
* 8. Pregnant or lactating women;
* 9. Patients with serious cardiovascular disease, uncontrollable infection, or other uncontrollable combined diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Ostomy reversal rate within 1 year after surgery | 1 year after surgery
  Ostomy reversal rate within 1 year after surgery
Incidence of anastomotic leakage within 6 months after surgery | 6 months after surgery
  Incidence of anastomotic leakage within 6 months after surgery

SECONDARY OUTCOMES:
Ostomy reversal rate within 2 years after surgery | 2 years after surgery
  Ostomy reversal rate within 2 years after surgery
Ostomy reversal rate within 3 years after surgery | 3 years after surgery
  Ostomy reversal rate within 3 years after surgery
Incidence of anastomotic leakage within 1 year after surgery | 1 year after surgery
  Incidence of anastomotic leakage within 1 year after surgery
Incidence of anastomotic leakage within 2 years after surgery | 2 years after surgery
  Incidence of anastomotic leakage within 2 years after surgery
Incidence of anastomotic leakage within 3 years after surgery | 3 years after surgery
  Incidence of anastomotic leakage within 3 years after surgery
Incidence of anastomotic stricture within 6 months after surgery | 6 months after surgery
  Incidence of anastomotic stricture within 6 months after surgery
Incidence of anastomotic stricture within 1 year after surgery | 1 year after surgery
  Incidence of anastomotic stricture within 1 year after surgery
Incidence of anastomotic stricture within 2 years after surgery | 2 years after surgery
  Incidence of anastomotic stricture within 2 years after surgery
Incidence of anastomotic stricture within 3 years after surgery | 3 years after surgery
  Incidence of anastomotic stricture within 3 years after surgery
Incidence of severe intestinal dysfunction at 1 year after ostomy reversal | 1 year after ostomy reversal
  Incidence of severe intestinal dysfunction at 1 year after ostomy reversal
Incidence of severe intestinal dysfunction at 2 years after ostomy reversal | 2 years after ostomy reversal
  Incidence of severe intestinal dysfunction at 2 years after ostomy reversal
Incidence of severe intestinal dysfunction at 3 years after ostomy reversal | 3 years after ostomy reversal
  Incidence of severe intestinal dysfunction at 3 years after ostomy reversal
Quality of life at 1 year after ostomy reversal | 1 year after ostomy reversal
  Quality of life at 1 year after ostomy reversal
Quality of life at 2 years after ostomy reversal | 2 years after ostomy reversal
  Quality of life at 2 years after ostomy reversal
Quality of life at 3 years after ostomy reversal | 3 years after ostomy reversal
  Quality of life at 3 years after ostomy reversal

REFERENCES:
- [Background] Delaney G, Jacob S, Featherstone C, Barton M. The role of radiotherapy in cancer treatment: estimating optimal utilization from a review of evidence-based clinical guidelines. Cancer. 2005 Sep 15;104(6):1129-37. doi: 10.1002/cncr.21324. PMID 16080176
- [Background] Andreyev J. Gastrointestinal symptoms after pelvic radiotherapy: a new understanding to improve management of symptomatic patients. Lancet Oncol. 2007 Nov;8(11):1007-17. doi: 10.1016/S1470-2045(07)70341-8. PMID 17976611
- [Background] Perrakis N, Athanassiou E, Vamvakopoulou D, Kyriazi M, Kappos H, Vamvakopoulos NC, Nomikos I. Practical approaches to effective management of intestinal radiation injury: benefit of resectional surgery. World J Gastroenterol. 2011 Sep 21;17(35):4013-6. doi: 10.3748/wjg.v17.i35.4013. PMID 22046090
- [Background] McCrone LF, Neary PM, Larkin J, McCormick P, Mehigan B. The surgical management of radiation proctopathy. Int J Colorectal Dis. 2017 Aug;32(8):1099-1108. doi: 10.1007/s00384-017-2803-y. Epub 2017 Apr 20. PMID 28429071
- [Background] Zhong Q, Yuan Z, Ma T, Wang H, Qin Q, Chu L, Wang J, Wang L. Restorative resection of radiation rectovaginal fistula can better relieve anorectal symptoms than colostomy only. World J Surg Oncol. 2017 Feb 2;15(1):37. doi: 10.1186/s12957-017-1100-0. PMID 28153025
- [Background] Meissner K. Late radiogenic small bowel damage: guidelines for the general surgeon. Dig Surg. 1999;16(3):169-74. doi: 10.1159/000018721. PMID 10436361
- [Background] Qin Q, Zhu Y, Wu P, Fan X, Huang Y, Huang B, Wang J, Wang L. Radiation-induced injury on surgical margins: a clue to anastomotic leakage after rectal-cancer resection with neoadjuvant chemoradiotherapy? Gastroenterol Rep (Oxf). 2019 Apr;7(2):98-106. doi: 10.1093/gastro/goy042. Epub 2018 Dec 11. PMID 30976422
- [Background] He Y, Zhou Z, Huang X, Guan Q, Qin Q, Zhu M, Wang H, Zhong Q, Chen D, Wang H, Fang L, Ma T. Laparoscopic Proximally Extended Colorectal Resection With Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Late Complications of Chronic Radiation Proctopathy. Front Surg. 2022 Apr 25;9:845148. doi: 10.3389/fsurg.2022.845148. eCollection 2022. PMID 35548188
- [Background] Anseline PF, Lavery IC, Fazio VW, Jagelman DG, Weakley FL. Radiation injury of the rectum: evaluation of surgical treatment. Ann Surg. 1981 Dec;194(6):716-24. doi: 10.1097/00000658-198112000-00010. PMID 7305485
- [Background] Jao SW, Beart RW Jr, Gunderson LL. Surgical treatment of radiation injuries of the colon and rectum. Am J Surg. 1986 Feb;151(2):272-7. doi: 10.1016/0002-9610(86)90086-3. PMID 3946764